CLINICAL TRIAL: NCT00419289
Title: Rehabilitation of COPD Patients: Can the Effect be Prolonged by Follow-up and Continued Rehabilitation
Brief Title: Optimizing the Effect of COPD Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KA20060179
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2007-01-08 (Estimated); Status verified 2007-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, rehabilitation, quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Behavioral: follow-up rehabilitation of participants with COPD

SUMMARY:
Patients with Chronic Obstructive Pulmonary Disease (COPD) may benefit from an 8-week pulmonary rehabilitation programme. However, the effect of the programme tends to attenuate with time. Patients who complete the programme are randomized to continued rehabilitation follow-up and control follow-up.

DETAILED DESCRIPTION:
Patients with Chronic Obstructive Pulmonary Disease (COPD) may benefit from an 8-week pulmonary rehabilitation programme according to guidelines of the Danish Society of Pulmonary Medicine. However, the effect of programme tends to attenuate with time. Patients who complete the programme are randomized to continued rehabilitation follow-up and control follow-up.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 < 60% of expected

Exclusion Criteria:

* Other severe chronic conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2007-01; Study Completion 2008-06

PRIMARY OUTCOMES:
Disease specific Quality of Life
Work Capacity

SECONDARY OUTCOMES:
Number of days admitted to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Vest, MD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Department of Internal Medicine M, Glostrup University Hospital, Copenhagen, Copenhagen, Denmark